CLINICAL TRIAL: NCT03327402
Title: A Phase 1 Open-label Study of the Safety, Tolerability, and Pharmacokinetics of d- and l-Amphetamine After Multiple Daily Doses of SHP465 6.25 mg Administered in Children Aged 4 to 5 Years With Attention-Deficit/Hyperactivity Disorder
Brief Title: Safety, Tolerability and Pharmacokinetics of SHP465 in Children Aged 4 to 5 Years With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP465-112
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: SHP465; ADHD; Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SHP465 (Experimental): Participants will receive SHP465 capsule at a dose of 6.25 mg, orally once daily for 4 weeks.
  Interventions: Drug: SHP465

INTERVENTIONS:
Drug: SHP465 — SHP465 capsule will be administered at a dose of 6.25 mg, orally once daily for 4 weeks. SHP465 is comprised of sulfate salts of dextroamphetamine and amphetamine, with dextroamphetamine saccharate and amphetamine aspartate monohydrate, which provide a composite enantiomer ratio of 3:1 d-amphetamine to l-amphetamine.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety, and tolerability of SHP465 in children aged 4 to 5 years with ADHD after multiple daily doses of 6.25 milligram (mg) SHP465

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 4-5 years inclusive at the time of consent with a primary diagnosis of ADHD (any subtype) based on a detailed psychiatric evaluation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) and has undergone nonpharmacological treatment or has a severe enough condition to consider enrollment without undergoing prior nonpharmacological treatment, based on the investigator's judgment or has never taken ADHD medication or has taken ADHD medication with unacceptable efficacy and/or tolerability.
2. Participant's parent/legally authorized representative (LAR) must sign the informed consent form, and there must be documentation of assent (if applicable) and is willing and able to fully comply with all of the testing and requirements defined in the protocol.
3. Participant during the screening period:

   i. Has a total score of ADHD-RS-5 >=28 for boys and >=24 for girls. ii. Has a Clinical Global Impressions-Severity of Illness (CGI-S) score >=4. iii.Functions at an age-appropriate level intellectually, as determined by the investigator.
4. Participant has the ability to take investigational product by either swallowing the capsule whole or sprinkling the capsule contents in applesauce and ingesting the entire mixture immediately without chewing.
5. Participant has lived with the same parent/LAR for at least 6 months.

Exclusion Criteria:

1. Prior enrollment or participation in the study.
2. Documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
3. Participant cannot swallow a pill and/or applesauce, or has an allergy to applesauce.
4. Participant is currently taking or has taken ADHD medication with acceptable efficacy and tolerability.
5. Participant has taken ADHD medication within 7 days prior to the administration of investigational product.
6. Participant has used any medication (including over-the-counter, herbal, or homeopathic preparations) within 30 days prior to the administration of investigational product or 5 half-lives, whichever is longer, with the exception of the following:

   i. Thyroid medication ii. Intermittent use of nonsteroidal anti-inflammatory drugs or acetaminophen iii. As needed use of a beta-agonists inhaler for mild asthma or exercise induced bronchospasm iv. Over-the-counter nonsedating antihistamines for allergies. v. Participant has continuously used oral corticosteroids >=7 days in 3 months prior to investigational product dosing. If continuous use was less than (<) 7 days, 1 month of washout prior to dosing of investigational product is required.
7. Within 30 days prior to the administration of investigational product (IP):

   i. Participant has used an IP.
   1. If the elimination half-life of the previous study's IP was less than 6 days, then the last dose of the previous IP should be 30 days prior to the first dose of SHP465.
   2. If the elimination half-life of the previous study's IP was greater than 6 days, then the last dose of the previous IP should be 5 half-lives prior to the dose of SHP465.
8. Glaucoma.
9. Known family history of sudden cardiac death or ventricular arrhythmia.
10. Known history of symptomatic cardiovascular disease, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, or other serious cardiac conditions placing them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
11. Any clinically significant ECG or clinically significant laboratory abnormalities at the first screening visit based on the investigator's judgment. A single retest of laboratory parameters is allowed based on the investigator's judgment.
12. Marfan's syndrome.
13. Blood pressure >= 95th percentile for age, sex, and height at the screening visit.
14. Height and weight <= 5th percentile for age and sex at the first screening visit.
15. Current abnormal thyroid function test results, defined as abnormal thyroid-stimulating hormone, thyroxine (T4), and tri-iodothyronine (T3) at the first screening visit. Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
16. History of seizures (other than infantile febrile seizures).
17. Current, controlled (requiring medication or therapy) or uncontrolled, comorbid psychiatric disorder including but not limited to any of the following comorbid Axis I disorders and Axis II disorders.
18. Currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of or is currently demonstrating active suicidal ideation.
19. History of physical, sexual, or emotional abuse.
20. Primary sleep disorder (eg, sleep apnea, narcolepsy).
21. Eating disorder.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- United States (8):
  - Preferred Research Partners, Little Rock, Arkansas
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - Qualmedica Research, LLC, Evansville, Indiana
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Pediatric Research Assn Inc, Dayton, Ohio
  - Professional Psychiatric Services (PPS), Mason, Ohio
  - Coastal Pediatric Associates, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions Inc, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ilic K, Kugler AR, Yan B, McNamara N. Pharmacokinetics, Safety, and Tolerability of SHP465 Mixed Amphetamine Salts After Administration of Multiple Daily Doses in Children Aged 4-5 Years with Attention-Deficit/Hyperactivity Disorder. CNS Drugs. 2022 Jan;36(1):71-81. doi: 10.1007/s40263-021-00870-5. Epub 2021 Nov 26. PMID 34826114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at eight centers in the United States between 13 March 2018 (first participant first visit) and 05 October 2018 (last participant last visit).
Pre-assignment Details: A total of 24 participants were enrolled and received the treatment. Of them 12 participants were included in the rich pharmacokinetic (PK) sampling group and 12 participants were included in the sparse PK sampling group. Overall, 22 participants completed the study.
Groups:
- SHP465: Participants aged 4-5 years received SHP465 capsule at a dose of 6.25 milligram (mg) orally once daily for 4 weeks.
Period: Overall Study
Arm/Group | SHP465
Started | 24
Rich PK Sampling Group | 12
Sparse PK Sampling Group | 12
Completed | 22
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other (Visit Out-Of-Window) | 1

BASELINE CHARACTERISTICS:
Population: Safety Set consisted of all enrolled participants who had taken at least one dose of investigational product.
Arm/Group | SHP465
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.8 (0.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Drug Concentration (Cmax) Occurred at the Time of Maximum Observed Concentration Sampled During a Dosing Interval (Tmax) of Plasma Dextroamphetamine (d-Amphetamine) and Plasma Levoamphetamine (l-Amphetamine)
Description: Maximum plasma drug concentration occurred at time of maximum observed concentration of plasma d-amphetamine and plasma l-amphetamine during a dosing interval were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: Pharmacokinetic (PK) set consisted of all participants in the safety set for whom at least one PK blood sample was collected. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Sparse PK sampling group were excluded from the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | SHP465
Number analyzed (Participants) | 11
nanogram per milliliter (ng/mL)
  d-Amphetamine | 31.37 (32.6)
  l-Amphetamine | 9.895 (34.7)

2. Primary Outcome: Trough Plasma Drug Concentration Ctrough at Steady State (Ctrough,ss) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Trough plasma drug concentration (predose concentrations collected at steady state) of plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Predose on Day 1 and Day 28 and at 24 hours (Day 29) postdose on Day 28
Population: PK set consisted of all participants in the safety set for whom at least one PK blood sample was collected. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Sparse PK sampling group were excluded from the PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
ng/mL
  d-Amphetamine | 7.934 (6.3077)
  l-Amphetamine | 3.092 (2.5253)

3. Primary Outcome: Time to Reach Maximum Observed Plasma Drug Concentration (Tmax) During Dosing Interval of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Time to reach maximum observed plasma drug concentration of plasma d-amphetamine and plasma l-amphetamine during a dosing interval were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: PK set consisted of all participants in the safety set for whom at least one post-dose PK blood sample was collected. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Sparse PK sampling group were excluded from the PK analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | SHP465
Number analyzed (Participants) | 11
hour
  d-Amphetamine | 7.917 [5.00 to 16.3]
  l-Amphetamine | 7.917 [5.00 to 16.3]

4. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero to the Last Timepoint (AUC0-t) During Sample Collection of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration-time curve from time zero to the last quantifiable concentration of plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | SHP465
Number analyzed (Participants) | 11
hour*nanogram per milliliter (hr*ng/mL)
  d-Amphetamine | 646.3 (27.5)
  l-Amphetamine | 222.1 (31.1)

5. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero Predose to Five Hours Postdose (AUC0-5) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration time curve from time zero predose to five hours postdose of plasma d-amphetamine and plasma d-amphetamine were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5 hours Postdose on Day 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
hr*ng/mL
  d-Amphetamine | 109.7 (36.1)
  l-Amphetamine | 34.53 (40.3)

6. Primary Outcome: Area Under the Concentration Time Curve From Time Five Hours to the Last Timepoint (AUC5-t) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration time curve from time five hours to the time of last quantifiable concentration of plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
hr*ng/mL
  d-Amphetamine | 549.9 (30.3)
  l-Amphetamine | 194.1 (34.1)

7. Primary Outcome: Area Under the Concentration-Time Curve From Time of Dosing to the Last Measurable Concentration (AUClast) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration-time curve from time of dosing to the last measurable concentration of plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
hr*ng/mL
  d-Amphetamine | 646.3 (27.5)
  l-Amphetamine | 222.1 (31.1)

8. Primary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval (24 Hours) at Steady State (AUCtau,ss) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration-time curve over the dosing interval (24 hours) at steady state of plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
hr*ng/mL
  d-Amphetamine | 520.6 (29.8)
  l-Amphetamine | 171.0 (32.9)

9. Primary Outcome: Terminal Rate Constant (Lambda z) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Terminal Rate Constant of plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: PK set consisted of all participants in the safety set for whom at least one PK blood sample was collected. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure at the specific categories. Sparse PK sampling group were excluded from the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | SHP465
Number analyzed (Participants) | 12
per hour
  d-Amphetamine: number analyzed (Participants) | 9
  d-Amphetamine | 0.06639 (15.5)
  l-Amphetamine: number analyzed (Participants) | 8
  l-Amphetamine | 0.05632 (15.3)

10. Primary Outcome: Total Body Clearance (CL/F) for Extravascular Administration of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Apparent total clearance of the plasma drug concentration of plasma d- amphetamine and plasma l-amphetamine after oral dose administration were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | SHP465
Number analyzed (Participants) | 11
Liter per hour (L/hr)
  d-Amphetamine | 5.618 (29.8)
  l-Amphetamine | 5.703 (32.9)

11. Primary Outcome: Terminal Half-life (t1/2) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Time required for the plasma drug concentration to reach half of its original value of plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | SHP465
Number analyzed (Participants) | 12
hour
  d-Amphetamine: number analyzed (Participants) | 9
  d-Amphetamine | 9.911 [8.42 to 14.1]
  l-Amphetamine: number analyzed (Participants) | 8
  l-Amphetamine | 12.16 [9.71 to 15.6]

12. Primary Outcome: Apparent Volume of Distribution (Vss/F) at Steady State of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Apparent volume of distribution at steady state of plasma d-amphetamine and plasma l-amphetamine after oral dose administration were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: Predose, 2, 5, 8, 12, 16, 24 hours (Day 8), 48 hours (Day 9) Postdose on Day 7
Population: PK set consisted of all participants in the safety set for whom at least one PK blood sample was collected.Here, number of participants analyzed signifies participants who were evaluable for this outcome measure at the specific categories. Sparse PK sampling group were excluded from the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | SHP465
Number analyzed (Participants) | 12
liter
  d-Amphetamine: number analyzed (Participants) | 9
  d-Amphetamine | 90.09 (34.3)
  l-Amphetamine: number analyzed (Participants) | 8
  l-Amphetamine | 109.4 (35.6)

13. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily had a causal relationship with this treatment. TEAEs was defined as AEs that start or deteriorate on or after the date of the first dose of investigational product (IP) and no later than 3 days following the last dose of IP.
Time Frame: From start of study drug administration up to follow-up (up to 5 weeks)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP465
Number analyzed (Participants) | 24
Participants | 11

14. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Reported as TEAEs
Description: Vital sign assessments included blood pressure, pulse, respiratory rate and body temperature. Any change in vital signs which were deemed clinically significant by the investigator were recorded as TEAE.
Time Frame: From start of study drug administration up to follow-up (up to 5 weeks)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP465
Number analyzed (Participants) | 24
Participants | 1

15. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Reported as TEAEs
Description: 12-lead ECG were evaluated. Any change in ECG assessments which are deemed clinically significant by the investigator were reported as TEAE.
Time Frame: From start of study drug administration up to follow-up (up to 5 weeks)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP465
Number analyzed (Participants) | 24
Participants | 0

16. Primary Outcome: Change From Baseline in Height at Final On-Treatment Assessment
Description: Height (in centimeters) was measured using a stadiometer with the participant standing on a flat surface without shoes and with the chin parallel to the floor. Final on-treatment assessment (FoTA) was defined as the last valid assessment obtained after baseline and while on IP (on or before 2 days after the last dose date).
Time Frame: FoTA (up to Day 30)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | SHP465
Number analyzed (Participants) | 22
centimeter (cm) | 1.601 (1.5073)

17. Primary Outcome: Change From Baseline in Weight at Final On-Treatment Assessment
Description: Weight (in kilograms) was measured using a calibrated scale. Participant should be in light clothes and without shoes. FoTA was defined as the last valid assessment obtained after baseline and while on IP (on or before 2 days after the last dose date).
Time Frame: FoTA (up to Day 30)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | SHP465
Number analyzed (Participants) | 24
kilogram (kg) | -0.305 (0.4268)

18. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Results Reported as TEAEs
Description: Clinical laboratory tests included biochemistry, endocrinology, hematology and urinalysis. Any change in clinical laboratory results which are deemed clinically significant by the investigator were reported as TEAE.
Time Frame: From start of study drug administration up to follow-up (up to 5 weeks)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP465
Number analyzed (Participants) | 24
Participants | 0

19. Primary Outcome: Number of Participants With Overall Quality of Sleep Assessed by Post Sleep Questionnaire (PSQ) at Final On-Treatment Assessment
Description: The PSQ was a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collected data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week. The assessment was done by the nature of the responses, not by a numbered scale. FoTA was defined as the last valid assessment obtained after baseline and while on IP (on or before 2 days after the last dose date).
Time Frame: FoTA (up to Day 30)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP465
Number analyzed (Participants) | 24
Participants
  FoTA: Overall quality of sleep - Very poor | 0
  FoTA: Overall quality of sleep - Poor | 4
  FoTA: Overall quality of sleep - Average | 6
  FoTA: Overall quality of sleep - Good | 11
  FoTA: Overall quality of sleep - Very Good | 3

20. Primary Outcome: Length of Time Awake Per Night Assessed by PSQ at Final On-Treatment Assessment
Description: The PSQ was a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collected data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week. FoTA was defined as the last valid assessment obtained after baseline and while on IP (on or before 2 days after the last dose date).
Time Frame: FoTA (up to Day 30)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SHP465
Number analyzed (Participants) | 14
minutes | 10.1 (9.86)

21. Primary Outcome: Length of Time to Fall Asleep Per Night Assessed by PSQ at Final On-Treatment Assessment
Description: as for outcome 20
Time Frame: FoTA (up to Day 30)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SHP465
Number analyzed (Participants) | 24
minutes | 19.8 (11.75)

22. Primary Outcome: Length of Time Sleeping Per Night Assessed by PSQ at Final On-Treatment Assessment
Description: as for outcome 20
Time Frame: FoTA (up to Day 30)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SHP465
Number analyzed (Participants) | 24
hours | 9.1 (1.41)

23. Primary Outcome: Total Sleep Disturbance Score of Children's Sleep Habits Questionnaire (CSHQ ) at Final On-Treatment Assessment
Description: The CSHQ was a validated, retrospective, parent-reported sleep screening tool. The questionnaire consisted of 35 items that yield a TSD score, as well as 8 subscale scores, including bedtime resistance, sleep duration, parasomnias, sleep disordered breathing, night wakings, daytime sleepiness, sleep anxiety, and sleep onset delay. Each item receives a score from 1 (meaning the problem occurs rarely) to 3 (meaning the problem usually occurs); therefore, a higher score is the worse outcome. Scale ranges are as follows: Bedtime Resistance: 6 to 18, Sleep Onset Delay: 1 to 3, Sleep Duration: 3 to 9, Sleep Anxiety: 4 to 12, Night Wakings: 3 to 9, Parasomnias: 7 to 21, Disordered Breathing: 3 to 9, Daytime Sleepiness: 8 to 24, and Total Disturbance (items from all scales): 33 to 99. A negative value indicated less sleep disturbance.
Time Frame: FoTA (up to Day 30)
Population: Safety set consisted of all enrolled participants who had taken at least one dose of investigational product. FoTA was defined as the last valid assessment obtained after baseline and while on IP (on or before 2 days after the last dose date).
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | SHP465
Number analyzed (Participants) | 24
Units on scale
  FoTA: Total Sleep Disturbance Score | 45.4 (8.21)
  FoTA: Bedtime Resistance | 10.1 (3.71)
  FoTA: Sleep Onset Delay | 1.4 (0.58)
  FoTA: Sleep Duration | 4.3 (1.68)
  FoTA: Sleep Anxiety | 6.2 (2.41)
  FoTA: Night Wakings | 4.1 (0.90)
  FoTA: Parasomnias | 8.9 (2.12)
  FoTA: Sleep Disordered Breathing | 3.2 (0.82)
  FoTA: Daytime Sleepiness | 10.6 (3.02)

24. Primary Outcome: Number of Participants With a Positive Response in Columbia-Suicide Severity Rating Scale (C-SSRS) at Final On-Treatment Assessment
Description: C-SSRS was a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts (suicidal ideation) and suicidal behaviors during the assessment period needed to be determine if a suicide-related thought or behavior were occurred. The assessment was done by the nature of the responses, not by a numbered scale. FoTA was defined as the last valid assessment obtained after baseline and while on IP (on or before 2 days after the last dose date).
Time Frame: FoTA (up to Day 30)
Population: Safety Set consisted of all enrolled participants who had taken at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP465
Number analyzed (Participants) | 24
Participants
  Suicidal Ideation | 0
  Suicidal Behavior | 0

25. Secondary Outcome: Observed Analyte Concentration at 12 Hours After Dose Administration (C12) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Observed analyte concentration of plasma d-amphetamine and plasma l-amphetamine at 12 hours after dose administration were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: 12 hours (Day 8) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
ng/mL
  d-Amphetamine | 24.59 (31.1)
  l-Amphetamine | 8.059 (33.2)

26. Secondary Outcome: Observed Analyte Concentration at 16 Hours After Dose Administration (C16) of Plasma d-Amphetamine and Plasma l- Amphetamine
Description: Observed analyte concentration of plasma d-amphetamine and plasma l-amphetamine at 16 hours after dose administration were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: 16 hours (Day 8) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
ng/mL
  d-Amphetamine | 20.53 (39.0)
  l-Amphetamine | 6.957 (40.7)

27. Secondary Outcome: Observed Analyte Concentration at 24 Hours After Dose Administration (C24) of Plasma d-Amphetamine and Plasma l- Amphetamine
Description: Observed analyte concentration of plasma d-amphetamine and plasma l-amphetamine at 24 hours after dose administration were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: 24 hours (Day 8) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
ng/mL
  d-Amphetamine | 11.16 (28.5)
  l-Amphetamine | 4.186 (32.7)

28. Secondary Outcome: Area Under the Concentration-Time Curve From Time Five Hours to Twelve Hours Postdose (AUC5-12) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration-time curve from time five hours to twelve hours postdose (AUC5-12) in plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method.Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: 5, 8, 12 hours Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
hr*ng/mL
  d-Amphetamine | 195.2 (32.6)
  l-Amphetamine | 61.88 (34.4)

29. Secondary Outcome: Area Under the Concentration-Time Curve From Time Twelve Hours to Sixteen Hours Postdose (AUC12-16) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration-time curve from time twelve hours to sixteen hours postdose (AUC12-16) in plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: 12, 16 hours Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
hr*ng/mL
  d-Amphetamine | 89.68 (31.7)
  l-Amphetamine | 29.92 (34.4)

30. Secondary Outcome: Area Under the Concentration-Time Curve From Time Sixteen Hours to Twenty-Four Hours Postdose (AUC16-24) of Plasma d-Amphetamine and Plasma l-Amphetamine
Description: Area under the concentration-time curve from time sixteen hours to twenty-four hours postdose (AUC16-24) in plasma d-amphetamine and plasma l-amphetamine were evaluated using rich sampling collection method. Values displayed do not necessarily reflect the actual precision obtained.
Time Frame: Week 4: 16, 24 hours (Day 8) Postdose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | SHP465
Number analyzed (Participants) | 11
hr*ng/mL
  d-Amphetamine | 122.1 (31.3)
  l-Amphetamine | 43.44 (34.0)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to 5 weeks)
Arm/Group | SHP465
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP465 (N=24)
Affect lability (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT03327402/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT03327402/SAP_001.pdf